CLINICAL TRIAL: NCT06612619
Title: Dyad Versus Single Instruction for Simulation-based Training in Proximal Femoral Fracture Osteosynthesis: a Non-inferiority Randomized Controlled Trial
Brief Title: Is Two-on-one Instruction in Virtual Reality Simulation-based Training of Operating Fractures of the Hip for Medical Students as Effective as One-on-one Instruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Amandus Gustafsson, Associate Professor, MD, PhD, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F-24056399
Record Dates: First submitted 2024-09-16; First posted 2024-09-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Learning Curves and Outcomes of Simulation-based Training
Keywords: Simulation-based training; Mastery standards; Proximal femoral fracture; Medical Education; Osteosynthesis; Orthopeadic surgery; Dyad instruction
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-on-one instruction to simulation-based training (No Intervention): The usual instruction with one instructor instructing the trainee in simulation-based training in osteosynthesis of proximal femoral fractures
- Dyad instruction (Active Comparator): Dyad or two-on-one instruction, where two trainees are instructed by an instructor at the same time and with the same time usage as in the non-intervention arm.
  Interventions: Behavioral: Dyad instruction

INTERVENTIONS:
Behavioral: Dyad instruction — Rather than being instructed solo or one-on-one the trainees are instructed in pairs of two (dyad).
  Arms: Dyad instruction

SUMMARY:
The training of orthopedic surgeons has historically relied heavily on an apprenticeship model as the primary way of teaching the various procedures an aspiring surgeon needs to master. However, due to work-hour restrictions, demand for operating room efficiency, lack of supervisors and a growing focus and concern for patient safety, this model is challenged. As the importance of proper education and supervision of surgeons in training is still monumental, simulation-based training (SBT) has gained popularity within most medical specialties, as it provides a safe, and realistic room for training, where surgeons can effectively enhance their operating technique without posing a threat to patient safety. Techniques within orthopedic surgery are no exception to this tendency, and several virtual reality simulators and SBT courses has been developed. This includes the well-established SBT course in proximal femoral fracture (PFF) osteosynthesis, where evidence supported mastery standards for antegrade nailing, dynamic hip screw, Hansson pins and canulated screws have been established. A course that is recommended in the national curriculum for Danish orthopedic surgeons in training.

This change into a more technology- and simulation-based training does however pose challenges, that needs to be acknowledged and addressed to ensure the quality of the education and clinical skills of the orthopedic surgeons.

A key challenge is the limited resource of qualified instructors. These instructors are mainly experienced surgeons with a demanding and busy schedule, who teach part time in addition to their clinical work. It has previously been shown that teaching skills are to be taught by doctors and that good clinicians are not automatically good educators. With the burden of a busy clinical schedule, these experienced surgeons have difficulties finding the time to learn teaching skills.

It can therefore be challenging to educate enough qualified instructors. This poses a rising concern as the field of SBT is only expected to grow, with more courses in continuous development. Thus, potentially limiting the accessibility to orthopedic SBT courses, including the PFF course.

A possible solution for this challenge is dyad introductions. By converting one-on-one introduction to SBT for trainees into one-on-two introduction, it is possible to double the number of participants getting introductions without increasing the teaching load or expenses. This could significantly reduce the needed faculty time per trainee. Several studies have shown beneficial learning outcomes of dyad training. However, it seems, that the positive effects of dyad training cannot be translated into all types of medical simulations, and some studies suggests that the complexity and nature of the simulation defines whether dyad training is beneficial . It is theorized, that the effect of dyad training is caused by the learning of motor skills through mirror neurons during observation, and the distribution of knowledge during complex simulations according to the cognitive load theory. This suggests, that dyad training may be most beneficial in complex simulations requiring high levels of motor skills such as complex surgical procedures.

To our knowledge, no studies exist that examines whether dyad introduction can be equally used in the simulations of orthopedic procedures in general or PFF surgery specifically.

The aim of this study was to examine whether dyad introduction is non-inferior to the current one-on- one student introduction.

ELIGIBILITY:
Inclusion Criteria:

* PGY 1 and 2 doctors working in an orthopeadic department

Exclusion Criteria:

* More than 10 osteosynthesis of proximal femoral fractures performed as the primary surgeon.
* Failure to achieve mastery within the 4-month follow-up window.s

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of two-hour self-trainin sessions to achieve mastery standard | From enrollment until mastery is achieved, or up to 4 months
  The embeeded test in the simulator has established mastery standards. The primary outcome is how many two hour training sessions the trainees has to attend to achieve the mastery standard

SECONDARY OUTCOMES:
Hands-on training time | From enrollment until mastery is achieved, or up to 4 months
  The hands-on time the trainee is actively training on the simulator
Test score of each iteration of training | From enrollment until mastery is achieved, or up to 4 months
  Test scores for each iteration of training until the trainee achieves the mastery standard
Failure to achieve mastery standard | Up to 4 months from enrollment
  Number of participants who do not achieve the mastery standard within 9 training sessions or within 4 months of enrollment (whichever comes first).
Calendar time to mastery | Up to 4 months from enrollment.
  Time from enrollment to achievement of the mastery standard within the 4-month follow-up period. Participants not achieving mastery within the window will be classified accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We will only share IPD based on a specific request or by demand of a journal